CLINICAL TRIAL: NCT04614194
Title: Single Cell Immune and Non-immune Correlates of Response to Neoadjuvant Abemaciclib and Letrozole in Hormone Receptor Positive Breast Cancer
Brief Title: Single Cell Immune and Non-immune Correlates of Response to Neoadjuvant Abemaciclib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Sangeetha Reddy, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2020-1043
Record Dates: First submitted 2020-10-13; First posted 2020-11-03 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Abemaciclib + Letrozole (Experimental): Patient will take twice daily abemaciclib and daily letrozole (Arm A) for 2 weeks prior to your planned standard treatment for breast cancer. In addition to tests and procedures that are part of your standard care, you will have a biopsy and blood draw for study purposes prior to starting study treatment.
  Interventions: Drug: Letrozole; Drug: Abemaciclib
- Arm B: Letrozole (Experimental): Patient will take daily letrozole only (Arm B) according to treatment arm for 2 weeks prior to your planned standard treatment for breast cancer. In addition to tests and procedures that are part of your standard care, you will have a biopsy and blood draw for study purposes prior to starting study treatment.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Oral. Tablets should be taken at the same times every day, with or without food.
Drug: Abemaciclib — Oral. Tablets should be taken at the same times every day, with or without food.
  Arms: Arm A: Abemaciclib + Letrozole

SUMMARY:
The purpose of this study is to better understand how the immune system plays a role in fighting breast cancer and specifically research if the immune system response against breast cancer can be improved with endocrine therapy and cyclin dependent kinase inhibitor therapy in patients with hormone receptor positive breast cancer. This will be studied by collecting tumor tissue and blood samples before and after 2 weeks of study treatment with commonly used endocrine therapy and cyclin dependent kinase inhibitor therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

* Clinical stage operable stage I, II, or III invasive mammary carcinoma, which is estrogen receptor or progesterone receptor positive by immunohistochemistry and HER2 negative by Herceptest (0 or 1+) or not amplified by in situ hybridization as per routine clinical testing.
* Have post-menopausal status, as defined by any of the following: Subjects at least 55 years of age OR Subjects under 55 years of age and amenorrheic for at least 12 months OR follicule stimulating hormone (FSH) values ≥ 40 IU/L and estradiol levels ≤ 40 pg/mL (140 pmol/L) or in postmenopausal ranges per local or institutional reference ranges.
* Breast tumor ≥1cm in diameter by either physical exam or ultrasound and suitable for pre and post-treatment tissue sampling.
* Meet either of 2 following criteria, for which neoadjuvant endocrine therapy for 2 weeks is deemed suitable: 1) disease that is planned for surgery as initial therapy, in which 2 weeks of neoadjuvant endocrine therapy is deemed suitable, 2) Disease for which neoadjuvant systemic therapy (either chemotherapy or endocrine therapy) may be planned, in which 2 weeks of neoadjuvant endocrine therapy prior to start of systemic therapy is deemed suitable.
* At least 18 years of age
* Performance status ECOG ≤ 2
* Have adequate organ function (ANC ≥1,500/mcL, Platelets ≥100,000/mcL, Hemoglobin ≥8 g/dL, Total bilirubin ≤1.5 × upper limit of normal, ALT and AST ≤3 × upper limit of normal, Creatinine clearance >30 mL/minute
* The patient is able to swallow oral medications
* Patients with a prior history of contralateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer.
* Women may have been taking tamoxifen or raloxifene as a preventive agent prior to study entry but must have discontinued the drug for at least 28 days prior to study enrollment.
* Subjects have ended hormone replacement therapy at least 7 days prior to receiving the first dose of randomized therapy.
* Ability to understand and the willingness to sign a written informed consent.
* A female of childbearing potential, must have a negative serum pregnancy test within 7 days of the first dose of abemaciclib and agree to use a highly effective contraception method during the treatment period and for 3 weeks following the last dose of abemaciclib. These criteria should not apply to most or all patients on the trial given the inclusion criteria is for post-menopausal patients only who should not be of childbearing potential.

Note: Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. Cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a patient or spouse/partner is determined to be pregnant following abemaciclib initiation, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation.

EXCLUSION CRITERIA:

* Active metastatic breast cancer, inflammatory breast cancer, or locally recurrent breast cancer.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
* Females who are pregnant, lactating, or premenopausal.
* Severe uncontrolled malabsorption condition or disease (i.e. grade 2 or higher diarrhea, severe malnutrition, short gut syndrome).
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Chemotherapy, radiotherapy, or any other cancer therapy for current diagnosis of breast cancer.
* Subjects may not have received or be receiving any other investigational agents for the treatment of the cancer under study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in T cell activation | After treatment ends (14 (+/- 3) days
  Change in T cell activation between matched pre-treatment and on-treatment tissue samples of responder patients treated with abemaciclib and letrozole. T cell activation will be defined as the density of granzyme positive CD8 T cells detected on multiplex immunohistochemistry. Responders are defined as having complete cell cycle arrest by Ki-67.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Reddy, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No